CLINICAL TRIAL: NCT06061952
Title: Prospective 12-week Randomized Controlled Trial (RCT) of Remotely- Delivered Customized Adherence Enhancement for Poorly Adherent Individuals With Schizophrenia (CAE-S) vs Enhanced Treatment as Usual (eTAU)
Brief Title: CAE for Poorly Adherent Individuals With Schizophrenia
Acronym: CAE-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Martha Sajatovic, Physician, UHMG, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY20230135
Record Dates: First submitted 2023-09-25; First posted 2023-09-29 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Customized Adherence Enhancement for Schizophrenia (CAE-S) (Experimental): CAE is an adjunctive (to standard medication treatment) behavioral intervention delivered virtually (real-time one on one video-conferencing) in 6 individual sessions. All participants will receive content from the 4 currently existing CAE modules delivered over a 6-session series spaced out over approximately 6-10 weeks. The material from the 4 modules will be broken down into predetermined sub-sections and delivered in 6 sessions. The modules themselves are delivered in sections (thematic units within the module) and do not correspond to a specific session. The 4 CAE modules are Psychoeducation, Communication with Providers, Medication Routines, and Substance Use.
  Interventions: Behavioral: Customized Adherence Enhancement for Schizophrenia (CAE-S)
- Enhanced Treatment as Usual (eTAU) (Other): To optimize control intervention rigor, the eTAU participants will view a pre-taped series of 6 videos (based on NAMI or DBSA general wellness guidelines) 1:1 with a therapist who has similar credentials and competency as the CAE mental health clinician. The therapist will view the video with the participant and field questions the patient may have.
  Interventions: Other: Enhanced Treatment as Usual (eTAU)

INTERVENTIONS:
Behavioral: Customized Adherence Enhancement for Schizophrenia (CAE-S) — 6-session series spaced out over approximately 6-10 weeks
  Arms: Customized Adherence Enhancement for Schizophrenia (CAE-S)
Other: Enhanced Treatment as Usual (eTAU) — eTAU participants will view a pre-taped series of 6 videos
  Arms: Enhanced Treatment as Usual (eTAU)

SUMMARY:
This project aims to evaluate the feasibility, acceptability and preliminary efficacy of remotely delivered CAE among patients with schizophrenia (CAE-S).

DETAILED DESCRIPTION:
Patients with schizophrenia will be randomly assigned to receive either CAE-S or eTAU following the baseline assessment. The primary feasibility outcomes will be attendance and patient satisfaction (Aim 1) and change from baseline to 12 weeks in schizophrenia symptoms as measured by the Positive and Negative Symptom Scale (PANSS) (Aim 2). An exploratory evaluation (Aim 3) will examine the posited mechanistic underpinnings of the CAE-S intervention by assessing change from screening to 12 weeks in psychotropic medication adherence as measured by the Tablets Routine Questionnaire (TRQ) and validated by eCAP (objective bottle openings). Secondary measures will include the Clinical Global Impression (CGI), functional status, quality of life and attitudes towards medication.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 18 and older with schizophrenia as confirmed by the Mini International Psychiatric Inventory (MINI)
* Prescribed an antipsychotic medication for treatment of schizophrenia
* Known to have medication treatment adherence problems as identified by the Tablets Routine Questionnaire (TRQ, 20% or more missed medications in past week or past month)
* Ability to be rated on psychiatric rating scales
* Currently in treatment or scheduled to receive treatment at a Community Mental Health Clinic (CMHC) or other clinical setting able to provide mental health care during and after study participation
* Able to provide written, informed consent to study participation
* Has access to electronic device and internet to complete sessions conducted on videoconferencing platform

Exclusion Criteria:

* Prior or current treatment with clozapine (clozapine therapy includes additional medication-related monitoring and clinical visits that may impact medication adherence)
* Medical condition or illness, which in the opinion of the research psychiatrist, would interfere with the patient's ability to participate in the trial
* Physical dependence on substances (alcohol or illicit drugs) likely to lead to withdrawal reaction during the course of the study in the clinical opinion of the treated research psychiatrist
* Immediate risk of harm to self or others
* Female who is currently pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-08-09 (Actual); Study Completion 2025-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Customized Adherence Enhancement for Schizophrenia (CAE-S) | Enhanced Treatment as Usual (eTAU)
Started | 19 | 17
Completed | 16 | 13
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Customized Adherence Enhancement for Schizophrenia (CAE-S) | Enhanced Treatment as Usual (eTAU) | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (10.9) | 47.4 (12.9) | 44.9 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 17 | 17 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 8 | 18
  Non-White | 9 | 9 | 18
Martial Status [Count of Participants; unit: Participants]
  Single, Never Married | 11 | 14 | 25
  Married | 4 | 0 | 4
  Previously Married (Separated/Divorced/Widowed) | 4 | 3 | 7
Years of Education [Mean (Standard Deviation); unit: years] | 13.4 (2.4) | 13.5 (2.2) | 13.4 (2.3)
Employment Status [Count of Participants; unit: Participants]
  Employed | 7 | 6 | 13
  Unemployed | 12 | 11 | 23
Health Insurance Status [Count of Participants; unit: Participants] — Participants may have more than 1 type of insurance, which is why the totals add up to more than the number of participants in a study arm.
  Participants
    Medicaid | 10 | 12 | 22
    Medicare | 9 | 9 | 18
    Private | 2 | 1 | 3
    No Insurance | 2 | 0 | 2
    Other | 1 | 0 | 1
Age at schizophrenia diagnosis [Mean (Standard Deviation); unit: years] | 23.8 (9.8) | 26.6 (8.3) | 25.1 (9.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.7 (5.3) | 33.6 (8.0) | 33.2 (6.6)
History of physical abuse [Count of Participants; unit: Participants] | 10 | 8 | 18
History of sexual abuse [Count of Participants; unit: Participants] | 9 | 7 | 16
PANSS total score [Mean (Standard Deviation); unit: units on a scale] — The PANSS is a clinician rated scale used for measuring symptom severity of patients with schizophrenia. Total scores range from 30 to 210, with higher scores indicating more severe schizophrenia.
  units on a scale | 61.7 (9.8) | 66.6 (8.5) | 64 (9.4)
Hospitalizations (lifetime) [Mean (Standard Deviation); unit: Number of hospitalizations] — Population: There were very few participants who had been hospitalized for substance use (4 participants overall - 3 in the CAE-S group and 1 in the eTAU group), so the decision was made to calculate mean number of hospitalizations using only those who had a hospitalization for substance use.
  Number of hospitalizations
    For schizophrenia | 6.7 (7.0) | 4.9 (3.3) | 5.6 (5.5)
    For substance abuse: number analyzed (Participants) | 3 | 1 | 4
    For substance abuse | 2.6 (1.2) | 3 — There was only 1 person in the eTAU group who had been hospitalized for substance abuse, therefore, a Standard Deviation cannot be calculated. | 2.8 (1)
Health resource use, past 3 months [Mean (Standard Deviation); unit: number of events]
  All-cause hospitalizations | 0.05 (0.2) | 0.24 (0.8) | 0.14 (0.5)
  Emergency room / urgent care | 1.3 (3.4) | 0.9 (1.2) | 1.1 (2.6)
  Any outpatient visits | 7.5 (9.6) | 6.4 (4.3) | 7 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Average Number of CAE-S Sessions Attended by Those in the CAE-S Group After 12 Weeks
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Number of sessions attended
Arm/Group | Customized Adherence Enhancement for Schizophrenia (CAE-S)
Number analyzed (Participants) | 19
Number of sessions attended | 4.89 (1.9)

2. Primary Outcome: Percentage of Subjects in the CAE-S Group That Agree or Strongly Agree That the Intervention Was Useful at 12 Weeks
Time Frame: 12 weeks
Population: Only 16 of the 19 participants randomized to CAE-S provided data on satisfaction with CAE-S
Measure: Number; unit: percentage of CAE-S participants
Arm/Group | Customized Adherence Enhancement for Schizophrenia (CAE-S)
Number analyzed (Participants) | 16
percentage of CAE-S participants | 93.8

3. Secondary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Total Score Between CAE-S and eTAU Groups at 12 Weeks
Description: The PANSS is a clinician rated scale used for measuring symptom severity of patients with schizophrenia. Total scores range from 30 to 210, with higher scores indicating more severe schizophrenia
Time Frame: 12 weeks
Population: Only 16 participants in the CAE-S group and only 13 participants in the eTAU group provided Week 12 data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Customized Adherence Enhancement for Schizophrenia (CAE-S) | Enhanced Treatment as Usual (eTAU)
Number analyzed (Participants) | 16 | 13
units on a scale
  Baseline | 60.9 (10.5) | 66.0 (9.7)
  Week 12 | 53.8 (9.0) | 54.2 (11.2)

4. Secondary Outcome: Change in Tablets Routine Questionnaire in the Past 7 Days (TRQ) at 12 Weeks
Description: The TRQ is a validated self-report measure that identifies proportion of days with missed doses in the past 7 days (past-week) and in the past 30 days (past-month). Lower scores (a smaller proportion/percentage n of missed medication) represent better adherence, while higher scores (a larger proportion/percentage of missed medication) represent worse adherence.
Time Frame: 12 weeks
Population: Only 16 participants in the CAE-S group and only 13 participants in the eTAU group provided Week 12 data
Measure: Mean (Standard Deviation); unit: Percentage of days with missed doses
Arm/Group | Customized Adherence Enhancement for Schizophrenia (CAE-S) | Enhanced Treatment as Usual (eTAU)
Number analyzed (Participants) | 16 | 13
Percentage of days with missed doses
  Baseline | 13.4 (16.5) | 13.2 (10.9)
  Week 12 | 17.9 (28.0) | 8.8 (11.0)

5. Secondary Outcome: Change in Tablets Routine Questionnaire in the Past 30 Days (TRQ) at 12 Weeks
Description: as for outcome 4
Time Frame: 12 weeks
Population: Only 16 participants in the CAE-S group and only 13 participants in the eTAU group provided Week 12 data
Measure: Mean (Standard Deviation); unit: Percentage of days with missed doses
Arm/Group | Customized Adherence Enhancement for Schizophrenia (CAE-S) | Enhanced Treatment as Usual (eTAU)
Number analyzed (Participants) | 16 | 13
Percentage of days with missed doses
  Baseline | 11.9 (20.7) | 7.7 (8.6)
  Week 12 | 7.4 (8.7) | 5.4 (7.0)

6. Secondary Outcome: Change in eCAP Use in the Past Week at 12 Weeks
Description: Study participants will be given an eCAP device for one of their pill bottles, which will record time/date of bottle opening. eCAP will be used to monitor the antipsychotic dosed most often (index drug). If more than one drug is dosed at the same frequency, the antipsychotic most recently added to the regimen will be the index drug.. Investigators will calculate a percent of doses taken by dividing the number of times the bottle is opened by the number of times it should have been opened as per the prescription.
Time Frame: 12 weeks
Population: We only have eCAP data on 11 participants in the CAE-S group and 8 participants in the eTAU group
Measure: Mean (Standard Deviation); unit: Percentage of missed doses
Arm/Group | Customized Adherence Enhancement for Schizophrenia (CAE-S) | Enhanced Treatment as Usual (eTAU)
Number analyzed (Participants) | 11 | 8
Percentage of missed doses
  Baseline | 20.8 (34.0) | 32.1 (32.2)
  Week 12 | 33.8 (36.9) | 50 (35.0)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Customized Adherence Enhancement for Schizophrenia (CAE-S) | Enhanced Treatment as Usual (eTAU)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/19 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Customized Adherence Enhancement for Schizophrenia (CAE-S) (N=19) | Enhanced Treatment as Usual (eTAU) (N=17)
Hospitalization due to pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization due to diabetes complications (Endocrine disorders) | 1 (1) | 0 (0)
Hospitalization due to renal complications (Renal and urinary disorders) | 1 (1) | 0 (0)
Hospitalization due to psychiatric symptoms (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT06061952/Prot_SAP_000.pdf